CLINICAL TRIAL: NCT01588210
Title: Fluoride Concentration in Inter-proximal Fluid From Dental Sealants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: WHO Collaborating Centre for Epidemiology and Community Dentistry (Unknown)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate professor of Community Dentistry, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120-01; 2011-10-11 (Registry Identifier: COMITATO DI BIOETICA DELLA ASL DI SASSARI)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Caries
Keywords: caries; sealant; fluoride; prevention; community dentistry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glass Ionomer Cement group (Experimental): a high-viscosity glass-ionomer cement (KETAC™ MOLAR APLICAP 3M Espe, Germany)
  Interventions: Other: Sealant application
- Resin Based Fluoride Group (Experimental): white photopolymerizable Resin-Based sealant containing fluoride (Helioseal F®, Ivoclar Vivadent AG, Fürstentum Liechtenstein)
  Interventions: Other: sealant application
- Resin Based sealant (Placebo Comparator): white photopolymerizable Resin-Based sealant (Concise 1930TM 3M Espe, Germany)
  Interventions: Other: sealant application

INTERVENTIONS:
Other: Sealant application — A high-viscosity glass-ionomer cement (KETAC™ MOLAR APLICAP 3M Espe, Germany) will be used.
  All sealants was applied following these steps: tooth isolation using cotton rolls or rubber dam; tooth cleaning using a rotary brush mounted on a low-speed contrangle with a prophylaxis pasta without fluoride; enamel etching using 37% phosphoric acid (H3PO4) for 30 seconds; rinse thoroughly with water and dry; placement a thin layer of sealant material and cure according to manufacturer's instructions and finally occlusion adjustment, if necessary.
  Arms: Glass Ionomer Cement group
Other: sealant application — A white photopolymerizable Resin-Based sealant containing fluoride (Helioseal F®, Ivoclar Vivadent AG, Fürstentum Liechtenstein) will be used.
  All sealants was applied following these steps: tooth isolation using cotton rolls or rubber dam (it was mandatory for both the RB sealants); tooth cleaning using a rotary brush mounted on a low-speed contrangle with a prophylaxis pasta without fluoride; enamel etching using 37% phosphoric acid (H3PO4) for 30 seconds; rinse thoroughly with water and dry; placement a thin layer of sealant material and cure according to manufacturer's instructions and finally occlusion adjustment, if necessary.
  Arms: Resin Based Fluoride Group
Other: sealant application — A white photopolymerizable Resin-Based sealant (Concise 1930TM 3M Espe, Germany) will be used.
  All sealants was applied following these steps: tooth isolation using cotton rolls or rubber dam (it was mandatory for both the RB sealants); tooth cleaning using a rotary brush mounted on a low-speed contrangle with a prophylaxis pasta without fluoride; enamel etching using 37% phosphoric acid (H3PO4) for 30 seconds; rinse thoroughly with water and dry; placement a thin layer of sealant material and cure according to manufacturer's instructions and finally occlusion adjustment, if necessary.
  Arms: Resin Based sealant

SUMMARY:
The hypothesis of this study is that the concentration of fluoride in oral interproximal fluids would increase more after using high-viscosity GIC as pit and fissure sealant, compared to Resin-Based sealants containing fluoride and RB sealants without fluoride content. To validate this hypothesis a randomized clinical trial was designed and performed in schoolchildren in order to evaluate fluoride release in inter-proximal fluid in vivo after the placement of three types of sealants: high-viscosity GIC, Resin-Based sealants containing fluoride and RB sealants without fluoride content.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are: year of birth between 2000 and 2002, informed consent signed by parents/guardians, presence of at least two permanent first molars completely erupted.

Exclusion Criteria:

* The exclusion criteria are: demineralized lesions and hypomineralized permanent molar, carious lesions or presence of filling on the occlusal surface of the first permanent molar, fixed orthodontic treatment.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2776 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Inter-proximal fluid fluoride concentration | 21 days after application
  Inter-proximal fluid was collected with a paper point in the mesial inter-proximal space of the sealed tooth for 15 seconds. Each sample was prepared for the analysis as follow: added of 0.5 ml TISAB III to reach a pH 5 and shaken with magnetic stirrer thermostated at 25°C for 15 seconds. 100 ml of the solution was then placed on a Petri dish for the analysis. Fluoride concentration was carried out with an Orion model 96.09 fluoride ion selective electrode and an Orion model 900200 double junction plastic body Ag/AgCl reference electrode with an Orion model 290 mV digital meter.

SECONDARY OUTCOMES:
caries incidence | 24 months
  measurement of tooth caries at D1, D2 D3 level (both enamel and dentinal caries)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Surgery, Microsurgery and Medicine Sciences University of Sassari, Sassari, Sardinia
  - WHO CC University of Milan, Milan

REFERENCES:
- [Derived] Cagetti MG, Carta G, Cocco F, Sale S, Congiu G, Mura A, Strohmenger L, Lingstrom P, Campus G; Italian Experimental Group on Oral Health. Effect of Fluoridated Sealants on Adjacent Tooth Surfaces: A 30-mo Randomized Clinical Trial. J Dent Res. 2014 Jul;93(7 Suppl):59S-65S. doi: 10.1177/0022034514535808. Epub 2014 May 20. PMID 24846910
- [Derived] Campus G, Carta G, Cagetti MG, Bossu M, Sale S, Cocco F, Conti G, Nardone M, Sanna G, Strohmenger L, Lingstrom P; Italian Experimental Group on Oral Health. Fluoride concentration from dental sealants: a randomized clinical trial. J Dent Res. 2013 Jul;92(7 Suppl):23S-8S. doi: 10.1177/0022034513484329. Epub 2013 May 20. PMID 23690357